CLINICAL TRIAL: NCT02785003
Title: Continuous Ketamine Infusion Versus Placebo in the Treatment of Acute Post-Surgical Pain: A Randomized Trial Evaluating the Efficacy of Ketamine in Colorectal Surgery
Brief Title: Ketamine in Colorectal Surgery
Acronym: KCRS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00027024
Record Dates: First submitted 2016-05-18; First posted 2016-05-27 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-05

CONDITIONS: Acute Pain; Pain, Postoperative; Colorectal Surgery
Keywords: Colorectal Surgery; Acute Pain; Pain; post-operative pain; ketamine
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Pain | interventions — Ketamine; Acetaminophen; Analgesics, Opioid; Opiate Alkaloids; Narcotics; Morphine; Hydromorphone; alvimopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine Infusion (Experimental): All infusion rates will be calculated based on ideal body weight. Patients will receive a bolus of the ketamine solution at a calculated dose of 0.25 mg/kg. A continuous infusion of ketamine will immediately follow at a rate of 2 mcg/kg/min. The continuous infusion to run for a duration of 48-hours.
  Interventions: Drug: Ketamine; Drug: Acetaminophen; Drug: Opioid; Drug: Alvimopan
- Saline Placebo (Placebo Comparator): All infusion rates will be calculated based on ideal body weight. Patients will receive a bolus of the saline solution at a calculated dose of 0.25 mg/kg. A continuous infusion of saline will immediately follow at a rate of 2 mcg/kg/min. The continuous infusion to run for a duration of 48-hours.
  Interventions: Drug: Placebo; Drug: Acetaminophen; Drug: Opioid; Drug: Alvimopan

INTERVENTIONS:
Drug: Placebo — Individuals enrolled into the control arm of the trial will receive a normal saline placebo infusion at a rate equivalent to the dosage of ketamine in the experimental arm.
  Other Names: NaCl Placebo Solution
  Arms: Saline Placebo
Drug: Ketamine — All individuals randomized to the experimental arm of the trial will receive ketamine therapy at a rate of 2 mcg/kg/hr dosed based on ideal body weight.
  Arms: Ketamine Infusion
Drug: Acetaminophen — All patients admitted to the hospital will be placed on scheduled acetaminophen 1000mg PO q 6 hours unless signs of liver disease/impairment or creatinine clearance < 35ml/min at which point dosage would be reduced to 650mg q 8 hours. Individuals unable to take oral medications would be placed on intravenous acetaminophen.
  Other Names: Tylenol
Drug: Opioid — All individuals will receive as needed opiate therapy as an adjunct to the scheduled medications and "ketamine/placebo" solution. Choice in opiate therapy will be at the discretion of the attending faculty. Dosage and adjustments will be in accordance with the institutional policy on appropriate opiate dosage adjustment.
  Other Names: Opiate, Narcotic; Morphine; Dilaudid
Drug: Alvimopan — All patients enrolled into the trial will be screened for eligibility for alvimopan utilization. Only in circumstances where patients are not on outpatient opioid medications and where they have not received any at time of arrival will alvimopan be administered. It will be given at least 30 minutes prior to surgery.
  Other Names: Entereg

SUMMARY:
This study will evaluate the effectiveness of ketamine infusions in the management of acute pain following open or laparoscopic colorectal surgery cases. Half of patients will receive the institutional standard of care and a placebo infusion (no active medication). The other half of patients will receive the institutional standard of care and a ketamine infusion. All subjects and staff will be blinded as to whether they are receiving placebo or ketamine.

DETAILED DESCRIPTION:
A prospective randomized, double blinded clinical trial of ketamine use in adult colorectal surgery patients will be conducted. The experimental arm of the trial will receive ketamine infusion therapy while the control arm of the trial receives saline placebo infusions at an equivalent rate. All patients enrolled into the trial will be enrolled in a standardized Enhanced Recovery after Surgery (ERAS) pathway which includes intravenous opioid medications for breakthrough pain, scheduled acetaminophen, and NSAIDs as indicated. All patients will be managed in accordance with the appropriate Division of Trauma and Acute Care Surgery and Division of Colorectal Surgery policies.

Potential participants will be screened at the time of outpatient clinic visits. Patients who require operative intervention for management of their colonic disease, both malignant and non-malignant, are eligible for enrollment. Individuals who present to the emergency department and are evaluated by the previously mentioned divisions will be screened for eligibility. If a potential participant qualifies for enrollment, he or she will be approached by one of the IRB approved study staff for consent. Prior to randomization and formal enrollment, an investigational drug services pharmacist will screen for any contraindication to potential ketamine therapy. Following investigator and pharmacy approval, patients will be randomized by the Investigational Drug Services (IDS). The two trial arms will be randomized in a 1:1 control to experimental fashion with randomization blocks conducted in sets of 4 patients.

Participants who are enrolled into the trial will undergo randomization into either the experimental or control arm by the IDS department at time of presentation to the hospital. The infusate will be prepared by the IDS department at a ketamine concentration of 500mg/250ml with all IV bags labeled "Investigational Ketamine / Placebo - PRO27024" prior to dispersal to the pre-operative nurse. All elective surgery patients will receive alvimopan beginning in the pre-operative area and administered by the RN at least 30 minutes prior to administration of narcotic medications. A total of 60 patients will be enrolled (see sample size calculation in c.2.3), 30 into each arm. All infusion rates will be calculated based on ideal body weight (IBW), unless actual body weight (ABW) is less than ideal. IBW is calculated for males as 50kg + 2.3*(number of inches over 5 feet) and for females as 45.5kg + 2.3*(number of inches over 5 feet). All investigational infusions will be started by the anesthesia resident or Certified Registered Nurse Anesthetists (CRNA) at the time of anesthesia induction. Patients will receive a bolus of the investigational solution at a calculated dose of 0.25 mg/kg over 5 minutes following anesthetic induction. A continuous infusion of the investigational solution will immediately follow at a rate of 2 mcg/kg/min. Timing of bolus administration along with time of initiation of continuous infusion will be documented with the continuous infusion to run for a duration of 48-hours.

All subjects will be assessed daily or more frequently for delirium. The institutional CAM and CAM-ICU Delirium screens, which have been validated in the literature, will be utilized (see appendices IV and V). Subjects may remove oneself from the trial or be un-blinded should he/she, pharmacy, and/or clinical staff deem it medically necessary. Medical necessity is determined by inability to treat without knowledge of trial assignment; otherwise treating staff will assume all patients have received ketamine. All adverse events will be recorded and if necessary subjects will be un-blinded in the event of a serious adverse event.

All adverse events will be recorded and if necessary subjects will be un-blinded in the event of a serious adverse event. The research team will monitor all study patients for any adverse event trends. Patients will be followed through the time of discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Surgical intervention required for the management of colonic disease
3. Admission to either the acute care surgery or colorectal surgery service with an anticipated inpatient hospital stay of 72 hours.

Exclusion Criteria:

1. History of adverse reaction to ketamine
2. Chronic opioid therapy for >3 weeks of >30mg oral morphine equivalents per day
3. Known substance abuse with prescription opioids or heroin
4. Anticipated post-operative intubation (>6hr duration)
5. History of psychosis
6. Active delirium
7. Glaucoma
8. Active acute coronary syndrome
9. Severe, poorly controlled hypertension (systolic blood pressure > 180)
10. Concurrent use of monoamine oxidase inhibitors (MAOIs)
11. Pregnancy
12. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Inpatient opiate consumption standardized to oral morphine equivalents. | 1st 48 hours post-infusion initiation
  Standardized to oral morphine equivalents

SECONDARY OUTCOMES:
Inpatient Opioid consumption standardized to oral morphine equivalents. | Duration of Hospitalization. Typical hospital duration for this patient population is 3-5 days.
  Standardized to oral morphine equivalents.
Opioid consumption standardized to oral morphine equivalents. | The 24-hours prior to leaving the hospital.
  Standardized to oral morphine equivalents. Will review opioid use in the 24-hours prior to the patient leaving the hospital.
AUCpain | 12-24 hours post infusion initiation
  Area under curve for the pain trajectory (AUCpain) during the 12 - 24 hours after initiation of pain treatment
AUCpain | 24-48 hours post-infusion initiation
  Area under curve for the pain trajectory (AUCpain) during the 24-48 hours after initiation of pain treatment
AUCpain | 6-12 hours post-infusion initiation
  Area under curve for the pain trajectory (AUCpain) during the 6-12 hours after initiation of pain treatment
Length of Stay | Participants will be followed for the duration of hospital stay, an expected average of 3-5 days.
  Participants will be followed from time of admission to time of discharge. The average hospital length of stay is expected to be 3-5 days.
ICU Length of Stay | Participants will be followed for the duration of hospital stay, an expected average of 3-5 days.
  Participants will be followed from time of admission to time of discharge. The average hospital length of stay is expected to be 3-5 days.
Opiate Side Effect Frequency | Participants will be followed for the duration of hospital stay, an expected average of 3-5 days.
  Nausea, Emesis, Pruritus, Sedation
Return of Bowel Function | Participants will be followed for the duration of hospital stay, an expected average of 3-5 days.
  Bowel Movements, Flatus

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Carver, MD, Principal Investigator — Medical College of Wisconsin; Carrie Y Peterson, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided